CLINICAL TRIAL: NCT04567797
Title: Assessing the Efficacy of Passive Exoskeletons for Construction Work: Lab-Based Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Xiang Yang, Principal Investigator, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007820207
Record Dates: First submitted 2020-09-04; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: passive exoskeleton

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Exoskeleton (Experimental): To compare the efficacy of four different exoskeleton devices, all participants will be asked to finish simulated construction tasks with each exoskeleton. Additionally, all participants will be asked to finish the same tasks without wearing an exoskeleton for reference.
  Interventions: Device: Laevo 2; Device: backX; Device: FLx ErgoSkeleton; Device: V22 ErgoSkeleton

INTERVENTIONS:
Device: Laevo 2 — The Laevo V2 is a wearable chest and back support exoskeleton. The Laevo transfers the from its chest pad to the thighs while bending forward. The passive exoskeleton (works with gas springs, not motors) transfers part of the load away from the back muscles, reducing the pressure on the spinal column. It provides a dampening effect on the back, reducing the risk of sudden back muscle contractions that needlessly overcompress the spine.
Device: backX — backX is a novel industrial exoskeleton that substantially augments its wearer and reduces the forces and torques on a wearer's lower back region (L5/S1 disc) by an average of 60% while the wearer is stooping, lifting objects, bending or reaching. backX augments the wearer's strength and can reduce the risk of back injuries among workers. It does not require external motors or power source. The mechanism of backX is similar to the first device "Laevo 2".
Device: FLx ErgoSkeleton — The FLx ErgoSkeleton is a range limiting work vest for physical work use. The FLx naturally reminds the user of the correct posture and lifting techniques while on the job site.
Device: V22 ErgoSkeleton — Similar to the FLx ErgoSkeleton, the V22 ErgoSkeleton keeps the position of the human body as to always stay within a safe body posture while lifting or moving heavy objects. The V22 ErgoSkeleton applies pressure to remind the user both during improper lifts and over rotation.
  In addition, the V22 ErgoSkeleton comes with two clutch controlled cables to assist in lifting and moving. The cables transfer part of the weight of the object being held directly to the V22 ErgoSkeleton vest, similar to other arm and shoulder support exoskeletons.

SUMMARY:
This project aims to assess the effectiveness and acceptability of four types of commercial Back support exoskeletons (BSEs) for concrete work tasks. BSEs are external wearable devices designed to reduce physical demands on the back by providing assistive moments to body joints to support muscles. There is considerable evidence to suggest such exoskeletons reduce the risks of back injuries for workers performing repetitive tasks. However, since the effects of using BSEs in concrete work tasks are still unknown, evidence-based information regarding effectiveness, productivity impact, and safety risks is required to help industries adopt BSEs as an ergonomic intervention.

DETAILED DESCRIPTION:
The experimental protocol will require approximately 3 hours of the participant's time. It will be comprised of six stages:

Stage I: Body Discomfort and Handedness Questionnaires First, the research team will administer an interview questionnaire to the participant to obtain information on participants' body pain/discomfort level and to determine the participant's hand dominance using the Edinburgh Handedness Inventory.

Stage II: Anthropometric body measurements and strength testing Several anthropometric body dimensions will be measured in the standing upright position using a standard tape measure and anthropometer. Body measurements will include standing height, shoulder height, waist to floor height, leg length, knee height, upper and lower arm length, foot length, and inter shoulder distance. Study participants' body weight will be measured using a standard weighing scale. Maximum power grip strength on both hands will be measured for 3 trials using a standard hand-held grip dynamometer.

Stage III: Fitting BSEs Four types of commercial BSEs (backX, Laevo 2, FLx ErgoSkeleton, V22 ErgoSkeleton) will be introduced to participants. Following manufacturers' instructions, participants will be allowed to test each device, fit the device to their body for comfort by using adjustable features (e.g., straps).

Stage IV: Optical motion capture marker, wearable inertial sensors, and surface electromyography (sEMG) sensor placement A commercial motion-capture system (Qualisys AB, Kvarnbergsgatan, Göteborg, Sweden) will be used to monitor and analyze body segment motion trajectories in a three-dimensional space. Several optical markers will be placed on anatomical landmarks of study participants including the head, shoulders, arms, hands, back, pelvis, legs, and feet. Hypo-allergenic double-sided tape will be used to attach the optical markers to the anatomical landmarks. Wearable inertial sensors will be attached using hypoallergenic double-sided tape at the low-back near the waist (S1), upper back (T6), sternum, upper arm (R, L), lower arm (R, L), thigh (R, L), and shank (R, L). Eight sEMG sensors will be placed on Descending Trapezius (TRP), Anterior Deltoid (AD), Iliocostalis Lumborum (ILL), Rectus Abdominis (RA), External Oblique (EO), Cervical Erector Spinae (CES), Latissimus Dorsi (LD), and Vastus Lateralis (VL) to measure muscle activation level while performing simulated work tasks, which are described in Stage VI.

Stage V: Maximum Voluntary Contraction (MVC) measurement for muscle activation While performing work tasks, muscle activation level varies between muscles and between subjects. A common way is to normalize myoelectric activities of each muscle for every participant by measuring isometric Maximal Voluntary Contraction (MVC). In this study, the investigators will measure 11 MVCs before the start of actual work tasks. Our MVC tests will be based on a study of trunk muscles. Before the MVC measurement, participants will be asked to warm up by 5 stretch exercises: (a) Stand upright with his feet shoulder-width apart. Place his hands on his buttocks for support. Look upwards and slowly lean backward. Keep his legs sturdy. (b) Stand upright with his feet shoulder-width apart. Place one hand on his buttocks for support. Look up and slowly lean backward. Reach over with his opposite hand. Rotate the upper body at the waist. (c) Kneel on one foot. Place his hands on his hips. Push hips forward. If necessary, hold on to something to keep balance. (d) Stand upright with his feet shoulder-width apart. Cross his arms and place his hands on shoulders. Slowly rotate his shoulders to one side. To increase the intensity of this stretch, use his hands to help rotate sideways. (e) Kneel on all fours. Support himself with one hand and reach towards his ankle with the other. Keep his back parallel to the ground. Keep the back straight, parallel to the ground, and his thigh in a vertical position. Distribute his weight evenly on both hands and knees. After the warm-up, the MVC testing will be performed, which includes (1) upper trunk flexion: subject will be in a sit-up posture positioned on a bench with the legs bent and feet strapped down with a belt. He then will attempt to flex the upper trunk in the sagittal plane while her thorax will be manually braced by the experimenter; (2) upper trunk twisting (R and L): In the same sitting supported position, the subject will attempt to twist the upper trunk in the horizontal plane while his thorax will be manually braced by the experimenter;(3) lower trunk flexion: subject will attempt to flex the lower trunk in the sagittal plane while he will be in a supine laying position, but with knees and hips both bent to approximately 90 degrees. His thorax will be strapped down with a belt and his legs will be manually braced by the experimenter; (4) lower trunk twisting (R and L): In the same lying and supported position, the subject will attempt to twist the lower trunk in the horizontal plane while his legs will be manually braced by the experimenter;(5) upper trunk bending (R and L): subject will attempt to side bend the upper trunk in the frontal plane while he will be in a side-lying position, with the knees bent and strapped with a belt, and thorax and arms will be manually braced by the experimenter; (6) lower trunk bending: subject will maintain a right and left side bridge position while maximally resisted downward pressure on the pelvis will be applied by the experimenter;(7) upper trunk extension: subject will be strapped in a prone position, with the torso horizontally cantilevered over the end of the bench (Biering-Sorensen position). He will then attempt to extend the upper trunk in the sagittal plane and retract the shoulders (squeezing the scapulae together) while manual resistance will be applied on the shoulders by the experimenter; (8) lower trunk extension: subject will attempt to extend the lower trunk and the hips against manual resistance when in a prone position, with the torso on the bench and the legs horizontally cantilevered over the end of the bench; (9) shoulder rotation and adduction (R and L): subject will attempt to adduct and internally rotate the shoulder against manual resistance with the shoulder abducted and elbow flexed, both to 90 degrees. In addition, two unresisted maximal abdominal contractions will be performed in standing; (10) maximal effort abdominal hollowing: subject will attempt to maximally activate the deep abdominal muscles while drawing in the lower abdomen; (11) maximal effort abdominal bracing: subject will attempt to maximally activate all the abdominal wall without any change in the position of the muscles. In all MVC testing, participants will be asked to exert their maximum force at a static posture (instructions will be given by our researcher) for every five seconds. For the first two seconds, they will be asked to ramp up to their maximum and maintain the force for the next three seconds. MVCs will be tested at least two times for each muscle group.

Stage VI: Data collection in simulated construction work tasks Postural data will be recorded from participants while performing six simulated concrete work tasks (i.e., shoveling, framing, carrying and lifting of construction materials, hammering, and tying rebars) at different intensities. The material they will be lifting, carrying, shoveling, and holding will not go over the safety limit of 30 lbs, as stated by NIOSH. Participants will perform the tasks with vs. without wearing different BSEs. Task trials will be video recorded for visual correspondence when analyzing motion capture and inertial sensor data. Participants will be given two minutes rest break between tasks and thirty seconds rest break between trials. The order of task conditions within each work task will be randomized.

* Task 1: Shoveling and moving construction material from location A to B. Distance between A and B will be set to 0.5m, both located at the ground level. Participants will be asked to shovel construction materials with three different weights (i.e., dirt, cement, and gravel). Participants will be asked to shovel at a high-frequency rate (15 scoops per minute).
* Task 2: Framing 30" wall using a power screwdriver. The frame will be placed on the floor, versus an elevated surface (28" height). Participants will be asked to use a power screwdriver to drive a screw into and out of the frame.
* Task 3: Carrying construction materials of different weights (i.e., wood frames and pipes) for up to 10 meters in each trial. The maximum weight of the carried materials will not exceed 30 lbs.
* Task 4: Lifting construction materials of different weights. The same materials will be used as the carrying task.
* Task 5: Pounding a punching bag located in the ground vs. 18 inches high vs. 36 inches high using a sledgehammer of different weights (i.e., 0, 6, 12, 16, and 20 lbs.).
* Task 6: Tying rebar in a framed grid located on different height levels (i.e., 0", 50").

The tasks and intensity levels were selected to be diverse yet reproducible (in terms of body postures) and resemble common tasks encountered in concrete work tasks.

Participants will be asked to answer questionnaires asking their experience, usability, and acceptability on each exoskeleton after they complete each work task.

The data collection process will end with removing optical markers and wearable sensors. Participants will be offered a rest break and refreshment if needed and followed by compensation and completing the payment form.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old.
* Be able to walk and/or lift heavy objects without pain/discomfort.

Exclusion Criteria:

* Have prior back/neck injuries or chronic pain in the last 6 months.
* Have a pacemakers.
* Have breast implants.
* Have removed the axillary lymph nodes.
* Pregnant women.
* Using blood thinning medications.
* Participants must consult a physician prior to participating this study if any of the following occurred before or during use: Inguinal hernia, hernia, knee injury hip/knee prosthesis, hyperextended knee, recent surgery, skin disease/injury, scars, inflammation, skin reddening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Muscle activities while performing simulated construction tasks | From admission to discharge, up to 3 hours
  Surface electromyography sensors will be placed on the following muscles of participants: Descending Trapezius (TRP), Anterior Deltoid (AD), Iliocostalis Lumborum (ILL), Rectus Abdominis (RA), External Oblique (EO), Cervical Erector Spinae (CES), Latissimus Dorsi (LD), and Vastus Lateralis (VL). Muscle activities while performing tasks represent the physical workload. Maximum Voluntary Contraction (MVC) technique will be used to normalize the muscle activities for comparison.
Body segment motions in a three-dimensional space measured by two methods | From admission to discharge, up to 3 hours
  Method 1: Wearable inertial sensors will be attached using hypoallergenic double-sided tape at the low-back near the waist (S1), upper back (T6), sternum, upper arm (R, L), lower arm (R, L), thigh (R, L), and shank (R, L). Body segment motions will be used to calculate relative angles, repetition count, duration of postures, which represent the physical workload of tasks.
  Method 2: Optical markers will be placed on anatomical landmarks of participants including the head, shoulders, arms, hands, back, pelvis, legs, and feet. The data collected my optical markers are mainly used for calibrating other sensors.

SECONDARY OUTCOMES:
Subjective review of workload level and experience using different exoskeleton | From admission to discharge, up to 3 hours
  Participants will be asked a set of subjective review questions on a questionnaire with eight sections:
  The difficulty of tasks: From "Very Difficult" to "Very Easy". "Easier" means a better outcome.
  Effectiveness: From "Very unhelpful" to "Very helpful". More helpful means a better outcome.
  Pain/discomfort level: From "Just noticeable" to "Intolerable" for different body locations. Less pain or discomfort means a better outcome.
  Acceptability: From "Very Uncomfortable" to "Very Comfortable". More comfortable means a better outcome.
  Fit/wearability by himself: From "Very difficult" to "Very easy". Easier means a better outcome.
  Preference of using this exoskeleton again and recommending to other people: From "Very unlikely" to "Very likely". More likely means a better outcome.
  An overall experience by ranking all exoskeletons: Options include 4 exoskeletons and "No exoskeleton". A higher rank means a better outcome.
  Open-ended interview.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Yang, Master, Principal Investigator — University of Arizona
Locations (1):
- Smart Life in Motion (SLIM) Lab, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to protect the privacy of participants.

REFERENCES:
- [Background] Vera-Garcia FJ, Moreside JM, McGill SM. MVC techniques to normalize trunk muscle EMG in healthy women. J Electromyogr Kinesiol. 2010 Feb;20(1):10-6. doi: 10.1016/j.jelekin.2009.03.010. PMID 19394867
- [Background] Axler CT, McGill SM. Low back loads over a variety of abdominal exercises: searching for the safest abdominal challenge. Med Sci Sports Exerc. 1997 Jun;29(6):804-11. doi: 10.1097/00005768-199706000-00011. PMID 9219209
- [Background] Juker D, McGill S, Kropf P, Steffen T. Quantitative intramuscular myoelectric activity of lumbar portions of psoas and the abdominal wall during a wide variety of tasks. Med Sci Sports Exerc. 1998 Feb;30(2):301-10. doi: 10.1097/00005768-199802000-00020. PMID 9502361
- [Background] Kavcic N, Grenier S, McGill SM. Quantifying tissue loads and spine stability while performing commonly prescribed low back stabilization exercises. Spine (Phila Pa 1976). 2004 Oct 15;29(20):2319-29. doi: 10.1097/01.brs.0000142222.62203.67. PMID 15480148
- [Background] Allison GT, Godfrey P, Robinson G. EMG signal amplitude assessment during abdominal bracing and hollowing. J Electromyogr Kinesiol. 1998 Feb;8(1):51-7. doi: 10.1016/s1050-6411(97)00004-7. PMID 9667034
- [Background] O'Sullivan PB, Twomey L, Allison GT. Altered abdominal muscle recruitment in patients with chronic back pain following a specific exercise intervention. J Orthop Sports Phys Ther. 1998 Feb;27(2):114-24. doi: 10.2519/jospt.1998.27.2.114. PMID 9475135
- [Background] Vera-Garcia FJ, Elvira JL, Brown SH, McGill SM. Effects of abdominal stabilization maneuvers on the control of spine motion and stability against sudden trunk perturbations. J Electromyogr Kinesiol. 2007 Oct;17(5):556-67. doi: 10.1016/j.jelekin.2006.07.004. Epub 2006 Sep 22. PMID 16996278
- [Background] Vera-Garcia FJ, Brown SH, Gray JR, McGill SM. Effects of different levels of torso coactivation on trunk muscular and kinematic responses to posteriorly applied sudden loads. Clin Biomech (Bristol). 2006 Jun;21(5):443-55. doi: 10.1016/j.clinbiomech.2005.12.006. Epub 2006 Jan 27. PMID 16442677
- [Background] Rogers, E. (2020). The Survey of Occupational Injuries and Illnesses Respondent Follow-Up Survey. Monthly Labor Review.
- [Background] Dong, X., Chowdhury, R., McCann, M., Trahan, C., & Gittle-man, J. S. (2008). The construction chart book: The US construction industry and its workers. In The Center for Construction Research and Training. Silver Spring.
- [Background] West GH, Dawson J, Teitelbaum C, Novello R, Hunting K, Welch LS. An analysis of permanent work disability among construction sheet metal workers. Am J Ind Med. 2016 Mar;59(3):186-95. doi: 10.1002/ajim.22545. Epub 2016 Jan 21. PMID 26792244
- [Background] Marcum J, Adams D. Work-related musculoskeletal disorder surveillance using the Washington state workers' compensation system: Recent declines and patterns by industry, 1999-2013. Am J Ind Med. 2017 May;60(5):457-471. doi: 10.1002/ajim.22708. Epub 2017 Mar 15. PMID 28295479
- [Background] Ngo, B. P., Yazdani, A., Carlan, N., & Wells, R. (2017). Lifting height as the dominant risk factor for low-back pain and loading during manual materials handling: A scoping review. IISE Transactions on Occupational Ergonomics and Human Factors, 5(3-4), 158-171.
- [Background] Kincl LD, Anton D, Hess JA, Weeks DL. Safety voice for ergonomics (SAVE) project: protocol for a workplace cluster-randomized controlled trial to reduce musculoskeletal disorders in masonry apprentices. BMC Public Health. 2016 Apr 27;16:362. doi: 10.1186/s12889-016-2989-x. PMID 27121123
- [Background] Dong, X., Betit, E., Dale, A., Barlet, G., and Wei, G. (2019). Trends of Musculoskeletal Disorders and Interventions in the Construction Industry. Quarterly Data Report by CPWR.
- [Background] Madinei S, Alemi MM, Kim S, Srinivasan D, Nussbaum MA. Biomechanical Evaluation of Passive Back-Support Exoskeletons in a Precision Manual Assembly Task: "Expected" Effects on Trunk Muscle Activity, Perceived Exertion, and Task Performance. Hum Factors. 2020 May;62(3):441-457. doi: 10.1177/0018720819890966. Epub 2020 Jan 14. PMID 31934773
- [Background] Alemi MM, Madinei S, Kim S, Srinivasan D, Nussbaum MA. Effects of Two Passive Back-Support Exoskeletons on Muscle Activity, Energy Expenditure, and Subjective Assessments During Repetitive Lifting. Hum Factors. 2020 May;62(3):458-474. doi: 10.1177/0018720819897669. Epub 2020 Feb 4. PMID 32017609
- [Background] Lim S, D'Souza C. Statistical prediction of load carriage mode and magnitude from inertial sensor derived gait kinematics. Appl Ergon. 2019 Apr;76:1-11. doi: 10.1016/j.apergo.2018.11.007. Epub 2018 Nov 29. PMID 30642513
- [Background] Lim S, D'Souza C. Statistical Prediction of Hand Force Exertion Levels in a Simulated Push Task using Posture Kinematics. Proc Hum Factors Ergon Soc Annu Meet. 2017 Sep;61(1):1031-1035. doi: 10.1177/1541931213601741. Epub 2017 Sep 28. PMID 29276370
- [Background] Lim S, D'Souza C. Inertial Sensor-based Measurement of Thoracic-Pelvic Coordination Predicts Hand-Load Levels in Two-handed Anterior Carry. Proc Hum Factors Ergon Soc Annu Meet. 2018 Sep;62(1):798-799. doi: 10.1177/1541931218621181. Epub 2018 Sep 27. No abstract available. PMID 32322142
- [Background] Lim, S. (2019). Combining Inertial Sensing and Predictive Modeling for Biomechanical Exposure Assessment in Specific Material Handling Work (Doctoral dissertation), University of Michigan, Ann Arbor.